CLINICAL TRIAL: NCT05864001
Title: STAR-C (Sustainable Behaviour Change for Health Supported by Person-Tailored, Adaptive, Risk-aware Digital Coaching in a Social Context) Digital Coaching Intervention
Brief Title: STAR-C Digital Coaching Intervention
Acronym: STAR-C
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-01461_Forte
Record Dates: First submitted 2023-04-05; First posted 2023-05-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-12

CONDITIONS: Healthy Lifestyle
Keywords: Prevention; Primary care; Digital intervention

STUDY DESIGN:
Intervention Model Description: One-sided crossover
Who Masked: Investigator
Masking Description: Upon their consent to participate in the study, baseline measurement will be conducted for each participant before their random allocation to different treatment arms. The research group will be blinded to the treatment assignment. The treatment assignment key will be revealed only after the intervention has been concluded and the analysis has been conducted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Immediate access to the digital coaching intervention
  Interventions: Behavioral: STAR-C mobile app
- Control (No Intervention): Delayed access to the digital coaching intervention, three months

INTERVENTIONS:
Behavioral: STAR-C mobile app — Digital coaching intervention for healthy lifestyle
  Arms: Intervention

SUMMARY:
Objectives: The overall objective is to evaluate the effectiveness of the STAR-C digital coaching intervention for health-related lifestyle behavioural change.

Study design: This intervention is designed as a two-arm individual pragmatic one-sided crossover randomised controlled trial, with participants receiving immediate access to the digital coaching intervention (Arm 1) and no digital coaching intervention (Arm 2, delayed access three months).

Setting: The intervention is integrated into the Västerbotten Intervention Programme (VIP) in Västerbotten Region. In total, 1000 participants will be recruited from all VIP-participating primary healthcare centres in Västerbotten, proportional to the size of the VIP participants in each centre. All participants will receive regular VIP intervention with the VIP nurse before recruitment into the STAR-C intervention study.

The intervention is planned to run for six months in total, with in-person recruitment at the baseline and follow-up at one, three, and six months. Individuals who are bedridden, terminally ill or have severe communication problems and those who receive behavioural change treatment at the Behavioural Medicine Clinic will be excluded.

Measures: The primary outcome of the intervention is change in the readiness for behaviour change at three months. The secondary outcomes include: (i) actual changes in the behaviours, including use of tobacco cessation clinics, higher smoking and snus cessation rate, reduction in alcohol consumption, adoption of healthy food habits, increased level of physical activity and reduction of sedentary behaviours, self-rated health and well-being, comparing baseline and follow-up data; (ii) patterns and usage of the digital tool during the intervention period (for the intervention group).

These outcomes will be measured quantitatively using questionnaires. In addition, interviews and group interviews will be conducted to explore the barriers and facilitators for the adoption and maintenance of the STAR-C digital coaching intervention for VIP nurses and the adult population.

DETAILED DESCRIPTION:
Objectives:

To evaluate the effectiveness of the STAR-C digital coaching intervention for health-related lifestyle behavioural change.

The specific objectives are to:

* Investigate to what extent STAR-C digital coaching intervention leads to change in the readiness for behavioural change (sub-study 1).
* Evaluate the effect of the digital intervention on behavioural change, including visit to tobacco cessation clinic, higher smoking and snus cessation rate, reduction in alcohol consumption, adoption of healthy food habits, increased level of physical activity and reduction of sedentary behaviours (sub-study 1).
* Evaluate the effect of the digital intervention on self-rated health and well-being (sub-study 1).
* Evaluate the cost-effectiveness of STAR-C digital coaching intervention compared to the existing VIP intervention in promoting behavioural change among the adult population (sub-study 2).
* Evaluate barriers and facilitators for adopting and maintaining the utilisation of STAR-C digital coaching intervention among the adult population (sub-study 3) and health professionals (sub-study 5).
* Evaluate barriers and facilitators for adopting and maintaining health-related lifestyle behavioural change among the adult population (sub-study 4).
* Analyse the different patterns of digital tool usage that could explain the effectiveness of the different behaviour change techniques embedded in the intervention and their relation to the participants and their characteristics (readiness for change, motivation, barriers, etc.), observed across age groups, gender, education level and geographical area of residence (sub-study 6).

Overall Study Design:

This is a two-arm individual pragmatic one-sided crossover randomised controlled trial conducted within the ongoing Västerbotten Intervention Programme (VIP) in Västerbotten Region in Sweden. VIP is integrated into primary care and invites inhabitants in Region Västerbotten to a health survey, including a comprehensive questionnaire and a systematic screening for cardiovascular risk factors, followed by a single individual health counselling with a trained nurse every ten years, at ages 40, 50, and 60 years. During the counselling, a "star profile" is used to illustrate the interrelationships between risk markers and behaviours and options for health promotion. All participants will receive the regular VIP intervention before recruitment to the study.

In intervention arm 1 (intervention arm), the participant will receive immediate access to digital coaching.

In intervention arm 2 (control arm), the participant will receive no digital coaching immediately but delayed access at three months.

Randomisation:

After completing the baseline assessment (a digital form), the application will automatically randomise the participants into one of the intervention arms. The investigators will use block randomisation to ensure a balanced number of participants recruited into the different arms in each intervention site.

Intervention:

The intervention embeds a set of behaviour change techniques:

* Goal setting for each domain of behaviour the participant wants to address
* Self-monitoring:

  * List of chosen activities relating to short and long-term goals for logging accomplishments
  * Visualisation of progress relating to particular selected behaviour(s) and the selected activities
  * Visualisation of overall status (STAR profile)
* Evidence/knowledge-based information and person-tailored advice, including information about health consequences
* Digital coach character with person-tailored behaviours to challenge and to support by providing reminders, feedback, and suggestions of goals, partly through text-based dialogues with the user.

Follow-up:

Follow-ups will be conducted at one, three, and six months. The application will send notifications two weeks before the follow-up time for the participants to fill in an online follow-up questionnaire as in the baseline. Three reminders will be sent to the participants, after a telephone survey will be conducted. In addition to the quantitative data, the investigators will also conduct qualitative studies.

Sample size:

A control prevalence of populations with readiness for behaviour change of 25% was assumed to yield a sample size of 328 participants in each arm that give 80% power at 95% confidence to detect a minimum of 40% increase (from 25% to 35%) in the prevalence of people with readiness for behaviour change in the intervention arm 1. After adjusting for a 50% oversample to allow for non-response, refusal or loss to follow-up, the investigators obtained the minimum sample size of 492 participants per arm, yielding a total of approximately 1000 participants being recruited into the trial.

Data analysis, sub-study 1 and 2:

Sub-study 1:

The investigators will use an intention-to-treat approach and assess differences in the groups using ANOVA and Chi-square tests for continuous and categorical variables, respectively. Longitudinal data using generalised estimating equations and mixed models will be used to assess the effect of time and the intervention on the outcomes. A latent transition analysis will be conducted to map different trajectories of readiness for behavioural change, comparing participants in the two arms.

Sub-study 2:

Costs for the development of the digital solution, the running costs for app maintenance, and costs for data storage in the server are regarded as fixed investment costs. The variable costs include costs for reimbursing the nurse's time spent in the initial training and time spent in implementing the intervention to the participants. When using a societal perspective in the analysis, the time used by the participants to participate in the intervention should also be accounted for as a cost. In the next step, the different costs are valued. In the valuation of various costs identified, the investigators will include costs from public material and the participants' time will be quantified with the opportunity cost approach. Alos, future savings will be related to reduced morbidity. The cost of developing the app will be measured by multiplying the estimated time by the current salaries. A first analysis relates the cost to the number of users. At the second step, the cost to users will be related to participants readiness to change their behaviours. A number of scenario-based cost effect analyses will be conducted, where published risk equations is used to draw conclusions. Another way to simplify the analysis is to calculate the number of gained quality-adjusted life years due to the intervention.

Summary of sub-studies 3-6:

Sub-study 3:

Aim: to explore the lived experience of using the STAR-C application among the adult population, including barriers and facilitators for use.

Sample: A sample of 8-10 STAR-C participants will be selected to represents a variation in age, gender, geographical location, and experience using digital tools.

Methods: The sub-study is based on ethnographic research methods. Personal photo/text journals and in-depth interviews will be used to explore the lived experience of using the STAR-C application, including barriers and facilitators for use. Study participants will be asked to document their use of the application visually and textually in a journal on three to five occasions (one week for each occasion), for six months. Visual and written journals allow individual participants to highlight matters they perceive to be important in long-term and day-to-day use of the application. Visual and textual journals will be complemented with in-depth interviews with study participants. In-depth interviews will allow participants to elaborate on matters identified and described in their visual and textual documentation, as well as for researchers to explore more specific matters related to participants' day-to-day use of the application, including barriers and facilitators for use. The study starts with an individual introduction where participants are informed about the purpose of the photo/text journal concerning their use of the STAR-C application. In-depth interviews will be conducted after three months of use of the application.

Analysis: The research material will be analysed using an ethnographic explorative approach based on Discourse theory and Science and Technology Studies.

Sub-study 4:

Aim: To understand the role of a digital tool in influencing health beliefs, readiness for change, and adoption of behavioural change.

Sample: Will be selected to represent a variation in geographical residence, age, gender, and experience of using digital tools.

The participants will be invited at 3 and 6 months after being included in the intervention, resulting in two rounds of interviews for those that agree upon this. Baseline data will be used as the foundation for the interview, where the participants will be asked to reflect upon the answers given at baseline. About 10-15 participants will be included in the study.

Methods: In-depth interviews will be used for the following study and if willing, interviewed at two occasions.

Analysis: In a deductive thematic analysis, the health belief model and the transtheoretical model of change will be used as frames of analysis.

Sub-study 5:

Aim: To explore healthcare professionals' experiences of using the STAR-C application as part of the VIP interventions, including perceptions of barriers and facilitators of using digital applications to help VIP participants to change and sustain health-related behaviours.

Sample: Approximately 15 healthcare professionals (nurses, assistant nurses, etc.) working with VIP will be selected based on having a variation in years of experience in working with the VIP, including health dialogues, and also experience in using digital tools for facilitating behavioural change. They will also represent a geographical variation.

Methods: The sub-study is based on group interviews with 15 participants, with 2-6 participants in each group interview. At least one group interview per the three broad geographical areas of the VIP will be conducted. The group interviews aim to identify pivotal matters connected to the overall aim of the sub-study. The sub-study will be conducted at least six months into the intervention so that staff have experience introducing and using the STAR-C application as part of the VIP.

Analysis: The research material will be analysed using Qualitative content analysis.

Sub-study 6:

Aim: To understand the role of the different behaviour change techniques embedded in the digital tool in influencing health beliefs, readiness for change and adoption of behavioural change, and other mechanisms of action, and how different participants utilise these for promoting healthy behaviour. Furthermore, the design and implementation of the behaviour change techniques will be further evaluated and refined, partly based on the participants' suggestions provided through the application.

Methods: Data collection is done using the STAR-C digital application. Data includes answers to questions, defined activities to meet goals, logging of activities, experienced effects of logged activities, sensor data counting steps, and logs of usage of different functionalities in the application.

Analysis: Quantitative analysis of use patterns and links between behaviour change techniques, mechanisms of action and domains of behaviour change. Ontological analysis of how participants define and adjust baby-step goals in the different domains of behaviour change. Qualitative analysis of open-ended questions embedded in the application using thematic analysis. Case studies of usage and behaviour change patterns over time.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Västerbotten Intervention Programme (VIP) who have received the VIP intervention.
* Has a smartphone.

Exclusion Criteria:

* Individuals who are bedridden, terminally ill, have severe vision/hearing problems, or with other hindrances to fulfilling the study protocol.
* Individuals who will be referred to the Behavioural medicine clinic (Beteendemedicin) for behavioural change treatment.

Ages: 39 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported readiness for behavioural change | 3 months
  The proportion of participants in different stages of behavioural change of (a) pre-contemplation; (b) contemplation; (c) preparation; (d) action; and (e) maintenance for different behaviours

SECONDARY OUTCOMES:
Change in tobacco habits | 3 months
  Self-reported change in use of tobacco products using questionnaire recommended by the Swedish National Board of Health and Welfare
Change in alcohol consumption | 3 months
  Self-reported change in alcohol consumption using questionnaire recommended by the Swedish National Board of Health and Welfare
Change in healthy food habits | 3 months
  Self-reported change of healthy food habits using questionnaire recommended by the Swedish Food Agency
Change in physical activity and sedentary behaviour | 3 months
  Self-reported change in level of physical activity and sedentary behaviours using questionnaire recommended by the Swedish National Board of Health and Welfare
Change in health-related quality of life | 3 months
  Self-reported health-related quality of life using the EQ-5D questionnaire
Change in well-being | 3 months
  Self-reported well-being using the World Health Organisation- Five (WHO-5) well-being questionnaire

OTHER OUTCOMES:
Costs | 3 months
  Cost-effectiveness evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Wennberg, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Primary health care, Region Västerbotten, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] Ng N, Eriksson M, Guerrero E, Gustafsson C, Kinsman J, Lindberg J, Lindgren H, Lindvall K, Lundgren AS, Lonnberg G, Sahlen KG, Santosa A, Richter Sundberg L, Weinehall L, Wennberg P. Sustainable Behavior Change for Health Supported by Person-Tailored, Adaptive, Risk-Aware Digital Coaching in a Social Context: Study Protocol for the STAR-C Research Programme. Front Public Health. 2021 Mar 1;9:593453. doi: 10.3389/fpubh.2021.593453. eCollection 2021. PMID 33732674

DOCUMENTS (2):
  • Study Protocol (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT05864001/Prot_002.pdf
  • Statistical Analysis Plan (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT05864001/SAP_003.pdf